CLINICAL TRIAL: NCT03697629
Title: A Phase 2 Open Label Study of an Accelerated Infusion Rate of Daratumumab in Patients With Relapsed and Refractory Multiple Myeloma
Brief Title: A Study of an Accelerated Infusion Rate of Daratumumab in Patients With Relapsed and Refractory Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Canadian Myeloma Research Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMRG 009
Record Dates: First submitted 2018-10-02; First posted 2018-10-05 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-02

CONDITIONS: Multiple Myeloma in Relapse
Keywords: Multiple Myeloma; Relapse; Refractory; Daratumumab; Accelerated Infusion
MeSH Terms: conditions — Multiple Myeloma; Recurrence | interventions — daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Daratumumab (Experimental): Increased infusion rate daratumumab monotherapy
  Interventions: Drug: Daratumumab

INTERVENTIONS:
Drug: Daratumumab — Patients will receive daratumumab, in the following schedule:
  Daratumumab 8mg/kg in 500 mL over 4 hours Cycle 1 Day 1, Daratumumab 16mg/kg in 500 mL over 90 minutes (20% of dose given in first 30 minutes and remaining 80% of dose given over 60 minutes) Cycle 1 Days 8, 15 and 22; Cycle 2 Days 1, 8, 15, and 22, and on Days 1 and 15 for Cycles 3-6.
  Other Names: Darzalex

SUMMARY:
Primary objective: To determine the incidence of infusion related reactions (IRR's) in the first 6 months of daratumumab administration.

DETAILED DESCRIPTION:
Study Design:

This is an open label phase II study of a daratumumab accelerated infusion regimen and a fixed pre- and post-medication regimen, in patients with relapsed and refractory Multiple Myeloma.

Patients will receive daratumumab, in the following schedule:

Daratumumab 8mg/kg in 500 mL over 4 hours Cycle 1 Day 1, Daratumumab 16mg/kg in 500 mL over 90 minutes (20% of dose given in first 30 minutes and remaining 80% of dose given over 60 minutes) Cycle 1 Days 8, 15 and 22; Cycle 2 Days 1, 8, 15, and 22, and on Days 1 and 15 for Cycles 3-6.

The study will begin with a 6-patient lead-in phase where safety with regards to the number of Grade 4 infusion related reactions with the accelerated infusion protocol will be evaluated in real time. Accrual to the study will not stop during this evaluation. The safety information obtained will be reviewed and evaluated in the context of previously published data. The review will be conducted by a 3-physician panel and if serious safety concerns (defined as Grade 4 infusion related reactions and/or death) are identified, the panel will make recommendations about protocol modifications if deemed necessary.

Pre- and post-medication regimen:

Montelukast 10 mg po x 2 days prior to daratumumab administration and 10 mg po the morning of daratumumab administration.

Cetirizine 10 mg po x 2 days prior to daratumumab administration and 10 mg po the morning of daratumumab administration.

Dexamethasone 20 mg on days of and day following daratumumab administration; starting Cycle 1 Day 15, dexamethasone 20 mg on day of daratumumab administration only.

Acetaminophen 975-1000 mg po 1 hour prior to daratumumab administration. Diphenhydramine 50mg IV 1 hour prior to daratumumab infusion.

Individual subjects will remain on treatment as long as there is no evidence of disease progression or unacceptable toxicity or until a patient/physician decision to discontinue is made. Disease assessments as determined by the Site Investigator will be made according to the IMWG response criteria guidelines for MM.1

As this study is designed to evaluate the IRRs associated with a shortened infusion time of daratumumab administration over a 6-month time period, subjects will be followed on study for a maximum of 6 months following enrollment. Following this time period, all subjects who continue to have a response to daratumumab will be taken off study. Although the study may end before subjects progress from their disease, daratumumab treatment will continue until disease progression in the absence of uncontrolled side effects or voluntary discontinuation of treatment for any reason, although drug will be supplied outside of the clinical trial setting.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females, age 18 years or older.
2. ECOG performance status score of 0, 1 or 2.
3. Life expectancy of at least 3 months
4. Measurable disease according to the IMWG criteria defined below (These baseline laboratory studies for determining eligibility must be obtained during the screening period within 28 days prior to start of study drug):

   1. Serum monoclonal paraprotein (M-protein) ≥ 10 g/L (if IgG) or ≥5g/L (if IgA, D, E or M).
   2. Urine M-protein ≥ 200 mg/24 h.
   3. Serum free light chains (FLC) assay: Involved FLC level ≥ 100 mg/L and an abnormal serum free light chain ratio (< 0.26 or > 1.65)
5. Received at least 3 prior lines of therapy including a proteasome inhibitor (≥2 cycles or 2 months of treatment) and an IMiD (≥2 cycles or 2 months of treatment) in any order or in combination during the course of treatment or subjects whose disease is double refractory to a PI and an IMiD. For subjects who have received more than 1 type of PI, their disease must be refractory to the most recent one. Similarly, for those who have received more than 1 type of IMID, their disease must be refractory to the most recent one.

   **A single line of therapy may consist of 1 or more agents, and may include induction, hematopoietic stem cell transplantation, and maintenance therapy (refer to Appendix 2). Radiotherapy, bisphosphonate, or a single short course of steroids (i.e. less than or equal to the equivalent of dexamethasone 40 mg/day for 4 days) would not be considered prior lines of therapy.
6. Have achieved at least a minimal response (MR) or better to at least one previous line of therapy as per IMWG response criteria.
7. The following laboratory results must be met within 10 days of first study drug administration:

   1. ANC ≥ 1.0 x 109/L
   2. Hemoglobin ≥ 80 g/L
   3. Platelets ≥ 70 x 109/L (or ≥50 x 109/L if ≥ 50% plasmacytosis in bone marrow)
   4. Calculated or measured CrCl ≥ 30 mL/min
   5. AST and ALT ≤ 3.0 x ULN
   6. Total bilirubin ≤ 2 x ULN unless known to have Gilbert's disease
   7. Corrected serum calcium ≤ 3.5 mmol/L
8. Have signed the informed consent documents indicating that the subject understands the purpose of the procedures required for the study and is willing to participate and adhere to the study protocol.
9. Females with child-bearing potential (FCBP†) must agree to use 2 reliable forms of contraception* simultaneously or practice complete abstinence from heterosexual contact for at least 28 days before starting study drug, while participating in the study (including during dose interruptions), and for at least 3 months after study treatment discontinuation.

   †Females of childbearing potential (FCBP): a female of childbearing potential is a sexually mature woman who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months).

   * The two methods of birth control used may be selected from the following categories, but the two methods cannot be selected from any one category: barrier method: i.e., condom (male or female) or diaphragm with spermicide; hormonal: i.e., contraceptive pill, patch; intrauterine device (IUD); vasectomy; or tubal ligation.
10. Females must agree to abstain from breastfeeding during study participation and 90 days after study drug discontinuation.
11. Males must agree to use a latex condom during any sexual contact with FCBP while participating in the study and for 3 months following discontinuation from this study, even if he has undergone a successful vasectomy.
12. Males must also agree to refrain from donating semen or sperm during the treatment phase and for 3 months after discontinuation from this study treatment.
13. All subjects must agree to refrain from donating blood while on study therapy and for 28 days after discontinuation from this study treatment.

Exclusion Criteria:

1. Prior exposure to daratumumab (or other anti-CD38 monoclonal antibody).
2. History of prior allogeneic stem cell transplantation and showing evidence of active graft-versus-host disease or graft-versus-host disease that requires immunosuppressive therapy.
3. Chemotherapy or other anti-myeloma therapy within 14 days prior to the first dose of study drug.
4. Treatment-related toxicity that has not recovered ≤Grade 1 unless deemed to be irreversible (an example of an irreversible toxicity would include steroid induced cataracts).
5. Subjects who have received steroids within 2 weeks prior to starting study treatment or who have not recovered from side effects of such therapy. Concomitant therapy medications that include corticosteroids are allowed if subject receive ≤ 10 mg of prednisone per day, or equivalent, as indicated for other medical conditions, or up to 100 mg of hydrocortisone as pre-medication for administration of certain medications or blood products prior to enrolment in this study.
6. Subjects who have received any investigational agents within 28 days or 5 half-lives (whichever is shorter, however the minimum allowed timeframe is 14 days) of the first dose (Cycle 1 Day 1).
7. Prior history of malignancies, other than MM, unless the subject has been free of the disease for 3 years or longer. Exceptions include the following:

   1. Basal or squamous cell carcinoma of the skin
   2. Carcinoma in situ of the cervix or breast
   3. Adenocarcinoma of the prostate (TNM stage of T1a or T1b)
8. Other concurrent severe and/or uncontrolled medical conditions (i.e. uncontrolled diabetes, active or uncontrolled infection, acute diffuse pulmonary disease, pericardial disease, uncontrolled thyroid dysfunction) including abnormal laboratory values, that could cause unacceptable safety risks or compromise compliance with the protocol.
9. Known chronic obstructive pulmonary disease (COPD), defined as a FEV1 < 50% predicted value.
10. Known moderate or severe persistent asthma within the last 2 years, or currently has uncontrolled asthma of any classification.
11. History of or current uncontrolled cardiovascular disease including:

    1. Unstable angina, myocardial infarction, or known congestive heart failure Class III/IV (Appendix 4) within the preceding 12 months
    2. Transient ischemic attack within the preceding 3 months, pulmonary embolism within the preceding 2 months.
    3. Any of the following: sustained ventricular tachycardia, ventricular fibrillation, Torsades de Pointes, cardiac arrest, Mobitz II second degree heart block or third-degree heart block; known presence of dilated, hypertrophic, or restrictive cardiomyopathy.
    4. QTc prolongation as confirmed by ECG assessment at screening (QTc >470 milliseconds).
12. Women who are pregnant, breastfeeding or planning to become pregnant while enrolled in this study, or within 6 months after the last dose of study medications. Male subject who plans to father a child while enrolled in this study, within 90 days after the last dose of study medications.
13. Subjects who are:

    1. Known seropositive for human immunodeficiency virus (HIV).
    2. Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (ie, subjects who are HBsAg negative but positive for antibodies to hepatitis B core antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination, do not need to be tested for HBV DNA by PCR.
    3. Seropositive for hepatitis C (except in the setting of a sustained virologic response [SVR], defined as aviremia at least 12 weeks after completion of antiviral therapy).
14. Known allergies, hypersensitivity to mannitol, corticosteroids, monoclonal antibodies or human proteins, or their excipients (refer to the Daratumumab PM), or known sensitivity to mammalian-derived products.
15. Known CNS involvement, amyloidosis, or currently active plasma cell leukemia.
16. Subjects who are receiving any other investigational agent.
17. Autologous, peripheral stem cell transplant within 12 weeks of the first dose of study drug.
18. Any other condition that, in the Investigator's opinion, would contraindicate the patient's participation in the clinical study due to safety concerns or compliance with clinical study procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-12-03 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Incidence of infusion related reactions (IRRs) | First 6 months of daratumumab administration
  For an accelerated infusion schedule compared to the approved schedule

SECONDARY OUTCOMES:
Overall response rate (ORR) | 6 months of daratumumab administration
  For this daratumumab dosing and infusion schedule according to IMWG criteria
Safety (adverse events) of study treatment | 6 months of daratumumab administration
  For this daratumumab dosing and infusion schedule, determine the incidence rates for adverse events using NCI CTCAE v5.0 grading. Generate a summary table for each term and body system, in addition to serious adverse events, subjects with related adverse events, subject deaths, and subjects who discontinue due to adverse events.

CONTACTS AND LOCATIONS:
Locations (6):
- Canada (6):
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - Hôpital Maisonneuve-Rosemont, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Hôpital de l'Enfant-Jésus, Québec, Quebec
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No